CLINICAL TRIAL: NCT00440505
Title: Effect of Nicotine on Chronic Pelvic Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Pamela Flood, Professor of Anesthesiology, Columbia University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAA4808
Record Dates: First submitted 2007-02-26; First posted 2007-02-27 (Estimated); Results first posted 2011-02-09 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-07

CONDITIONS: Pelvic Pain
Keywords: chronic pain; pelvic pain; nicotine patch
MeSH Terms: conditions — Pelvic Pain; Chronic Pain | interventions — Nicotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Subjects applied a placebo patch (0 mg) in the morning and removed it at bedtime for one day.
  Interventions: Drug: Placebo
- Nicotine (5 mg) (Experimental): Subjects applied a nicotine patch (5 mg) in the morning and removed it at bedtime for one day.
  Interventions: Drug: Nicotine (5 mg)
- Nicotine (10 mg) (Experimental): Subjects applied a nicotine patch (10 mg) in the morning and removed it at bedtime for one day.
  Interventions: Drug: Nicotine (10 mg)

INTERVENTIONS:
Drug: Placebo — Subjects applied a placebo patch (0 mg) in the morning and removed it at bedtime for one day.
  Arms: Placebo
Drug: Nicotine (5 mg) — Subjects applied a nicotine patch (5 mg) in the morning and removed it at bedtime for one day.
  Arms: Nicotine (5 mg)
Drug: Nicotine (10 mg) — Subjects applied a nicotine patch (10 mg) in the morning and removed it at bedtime for one day.
  Arms: Nicotine (10 mg)

SUMMARY:
The purpose of this study is to test whether transdermal nicotine reduces pain among women with chronic pelvic pain.

DETAILED DESCRIPTION:
Potential subjects are female non-smokers presenting to their physicians for treatment of chronic pelvic pain. When consented, the subjects fill out a questionnaire on demographic information and pain experience. The trial is conducted at home over three days. Each subject uses three different levels of nicotine (0mg, 5mg, and 10mg) administered in a random order; the study is double-blinded and patients act as their own controls. Subjects apply the placebo or nicotine patches in the morning and remove them in the evening when they fill out a pain diary for the day. During the study, patients will continue their typical course of pain medication and report pain medication use in the pain diary.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pelvic pain
* Aged 18-60 years
* Female

Exclusion Criteria:

* Uncontrolled hypertension
* Cardiovascular disease
* Current analgesic abuse
* Pregnancy
* Current usage of nicotine patch or gum
* Allergy to adhesive tape

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2004-02; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Flood, MD, Principal Investigator — Columbia University; Jessamyn Conell-Price, BA, Study Director — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This double-blind prospective study was approved by the Institutional Review Board of Columbia University Medical Center. Written consent was obtained from all subjects. Women presenting with chronic pelvic pain to a gynecologist or to the pain clinic at New York Presbyterian Hospital were eligible for inclusion.
Pre-assignment Details: Twenty-six women were recruited for the study. Six women declined to participate after consenting but before commencing treatment; these women are not included in the analysis.
Groups:
- Placebo First, Then Nicotine 5 mg, Then Nicotine 10 mg: Placebo patch for one day in first intervention period, nicotine 5 mg patch for one day in second intervention period and nicotine 10 mg patch for one day in the third intervention period.
- Placebo First, Then Nicotine 10 mg, Then Nicotine 5 mg: Placebo patch for one day in first intervention period, nicotine 10 mg patch for one day in second intervention period and nicotine 5 mg patch for one day in the third intervention period.
- Nicotine 5 mg First, Then Nicotine 10 mg, Then Placebo: Nicotine 5 mg patch for one day in first intervention period, nicotine 10 mg patch for one day in second intervention period and placebo patch for one day in the third intervention period.
- Nicotine 5 mg First, Then Placebo, Then Nicotine 10 mg: Nicotine 5 mg patch for one day in first intervention period, placebo patch for one day in second intervention period and nicotine 10 mg patch for one day in the third intervention period.
- Nicotine 10 mg First, Then Nicotine 5 mg, Then Placebo: Nicotine 10 mg patch for one day in first intervention period, nicotine 5 mg patch for one day in second intervention period and placebo patch for one day in the third intervention period.
- Nicotine 10 mg First, Then Placebo, Then Nicotine 5 mg: Nicotine 10 mg patch for one day in first intervention period, placebo patch for one day in second intervention period and nicotine 5 mg patch for one day in the third intervention period.
Period: First Intervention
Arm/Group | Placebo First, Then Nicotine 5 mg, Then Nicotine 10 mg | Placebo First, Then Nicotine 10 mg, Then Nicotine 5 mg | Nicotine 5 mg First, Then Nicotine 10 mg, Then Placebo | Nicotine 5 mg First, Then Placebo, Then Nicotine 10 mg | Nicotine 10 mg First, Then Nicotine 5 mg, Then Placebo | Nicotine 10 mg First, Then Placebo, Then Nicotine 5 mg
Started | 5 | 2 | 1 | 2 | 5 | 5
Completed | 5 | 2 | 1 | 2 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention
Arm/Group | Placebo First, Then Nicotine 5 mg, Then Nicotine 10 mg | Placebo First, Then Nicotine 10 mg, Then Nicotine 5 mg | Nicotine 5 mg First, Then Nicotine 10 mg, Then Placebo | Nicotine 5 mg First, Then Placebo, Then Nicotine 10 mg | Nicotine 10 mg First, Then Nicotine 5 mg, Then Placebo | Nicotine 10 mg First, Then Placebo, Then Nicotine 5 mg
Started | 5 | 2 | 1 | 2 | 5 | 5
Completed | 5 | 2 | 1 | 2 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention
Arm/Group | Placebo First, Then Nicotine 5 mg, Then Nicotine 10 mg | Placebo First, Then Nicotine 10 mg, Then Nicotine 5 mg | Nicotine 5 mg First, Then Nicotine 10 mg, Then Placebo | Nicotine 5 mg First, Then Placebo, Then Nicotine 10 mg | Nicotine 10 mg First, Then Nicotine 5 mg, Then Placebo | Nicotine 10 mg First, Then Placebo, Then Nicotine 5 mg
Started | 5 | 2 | 1 | 2 | 5 | 5
Completed | 5 | 2 | 1 | 1 | 5 | 5
Not Completed | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Entire Study Population
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Pain Score
Description: Pain assessment by patient reported in visual analog score (VAS) with 0=no pain and 10=worst pain.
Time Frame: 1 day
Population: This analysis was per protocol. One patient dropped out of the study before the third intervention period. This patient does not have data for the 10 mg nicotine patch.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Placebo: Placebo patch administered for one day in either first intervention period, second intervention period or third intervention period.
- Nicotine 5 mg: Nicotine 5 mg patch administered for one day in either first intervention period, second intervention period or third intervention period.
- Nicotine 10 mg: Nicotine 10 mg patch administered for one day in either first intervention period, second intervention period or third intervention period.
Arm/Group | Placebo | Nicotine 5 mg | Nicotine 10 mg
Number analyzed (Participants) | 20 | 20 | 19
Units on a scale | 7.1 (3.1) | 6.4 (3.0) | 6.9 (3.2)

2. Secondary Outcome: Patient Self-assessment of Psychological Distress
Description: Patient self-assessment of psychological distress in brief rating scale with no psychological distress=0 and maximum psychological distress=90.
Time Frame: 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Nicotine 5 mg | Nicotine 10 mg
Number analyzed (Participants) | 20 | 20 | 19
Units on a scale | 40.2 (18.3) | 36.7 (18.6) | 37.5 (18.2)

3. Secondary Outcome: Number of Participants Who Reported an Increase in Daily Pain Medication Regime
Description: Number of participants who reported increases in daily pain medication after treatment with each intervention compared to their normal daily pain medication regime.
Time Frame: 1 day
Population: This analysis was per protocol. Only data from those patients who returned the pain diaries with the above information to the research staff by mail were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Placebo | Nicotine 5 mg | Nicotine 10 mg
Number analyzed (Participants) | 13 | 13 | 13
Participants | 2 | 3 | 2

4. Secondary Outcome: Nausea
Description: Nausea assessment by patient reported on a numerical rating scale (NRS) with 0=no nausea and 10=extreme nausea.
Time Frame: 1 day
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Nicotine 5 mg | Nicotine 10 mg
Number analyzed (Participants) | 13 | 13 | 13
Units on a scale | 2.3 (1.8) | 2.3 (2.1) | 2.3 (2.1)

ADVERSE EVENTS:
Groups:
- Placebo: Non-smokers with the placebo patch
- Nicotine 5mg: Non-smokers with the Nicotine 5mg patch
- Nicotine 10mg: Non-smokers with the Nicotine 10mg patch
Arm/Group | Placebo | Nicotine 5mg | Nicotine 10mg
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes